CLINICAL TRIAL: NCT05498467
Title: The Role of Interleukin-1 Beta Targeted Therapy for Patients Suffering From Allergic Contact Dermatitis: A Randomized Controlled Trial With Anakinra vs. Placebo
Brief Title: The Role of Interleukin-1 Beta Targeted Therapy for Patients Suffering From Allergic Contact Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Kelvin Yeung, MD, Principal Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEOSIC
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anakinra (Active Comparator)
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium Chloride 9mg/ml Injection

INTERVENTIONS:
Drug: Anakinra — 100 mg Anakinra injections s.c.
  Arms: Anakinra
Drug: Sodium Chloride 9mg/ml Injection — 9 mg Sodium Chloride injections s.c.
  Arms: Placebo

SUMMARY:
The study will investigate if Anakinra can ameliorate allergic contact dermatitis in participants with known nickel allergy

ELIGIBILITY:
Inclusion Criteria:

* Aged at least eighteen years old.
* Able to provide written informed consent.
* Have a medical diagnosis of nickel allergy with at least a +2 reaction on the
* ICDRG scoring system when challenged with nickel.
* Fitzpatrick skin type 1-4.
* Able to speak and understand Danish.

Exclusion Criteria:

* Received any topical immunomodulating or immunosuppresive treatment on the lower back two weeks prior, or applied crème/lotion on the lower back 24 hours prior to day 0.
* Received systemic immunomodulating or immunosuppressive treatment four weeks prior to day 0.
* Any skin lesions at the area of interest such as nevi, scar tissue or pigment changes.
* Dermatitis and/or infection.
* Recent (3 months or less) administration of a live virus vaccine.
* Women of childbearing potential who are not taking adequate contraception or who are pregnant, plan to become pregnant during the study duration or lactating.
* Taking part in any other intervention study.
* Has any other condition which would, in the Investigator's opinion, deem the patient unsuitable for participation in the study (e.g. condition requiring long term or frequent oral steroid use).
* Presence of any condition or use of any medication which precludes the use of the study drug.
* Allergy to any of the ingredients in the drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Placebo | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.1) | 36.6 (13.4) | 38.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Clinical Reaction
Description: Number of participants with a lower clinical ICDRGscoring in the active treatment group compared to placebo
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 9 mg Sodium Chloride injections s.c.
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 12 | 8
Participants
  Clinical treatment effect | 0 | 0
  No clinical treatment effect | 12 | 8

ADVERSE EVENTS:
Time Frame: through study completion (45 days)
Description: Adverse events were collected at each visit.
Arm/Group | Anakinra | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT05498467/Prot_SAP_000.pdf